CLINICAL TRIAL: NCT01574040
Title: A Before-and-after Study to Evaluate Effects of Low-cost Interventions for Promoting Healthy Lifestyle Modifications
Brief Title: The Lifestyle moDIfCation Study
Acronym: LUDIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, dr.Frank L.J. Visseren, Professor of Vascular Medicine, Internist, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Vasc-UMCU-14B
Record Dates: First submitted 2012-02-09; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Lifestyle; Lifestyle modification; Behavior; Primary prevention; Healthy staff and visitors of an Academic Hospital
MeSH Terms: conditions — Behavior | interventions — Margarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Staff (and visitors) of the University Medical Centre Utrecht (Experimental): This is a dynamic study population
  Interventions: Behavioral: Promotion of stair climbing; Behavioral: Promotion of a low-salt soup alternative for the 'soup of the day'; Behavioral: Promotion of a low-fat alternative for the butter croissants; Behavioral: Exchange of the basket positions of butter and margarine in the UMC staff restaurant between convenient and harder to reach locations

INTERVENTIONS:
Behavioral: Promotion of stair climbing — Application of labels on all UMC elevator doors stating: " If you take the stairs, you will burn 11 times more calories."
Behavioral: Promotion of a low-salt soup alternative for the 'soup of the day' — Promotion of a low-salt soup alternative for the 'soup of the day' in the UMC staff restaurant, using a sign stating: "The cream soup contains 30% less salt and contributes to a healthy blood pressure."
Behavioral: Promotion of a low-fat alternative for the butter croissants — Promotion of a low-fat alternative for the butter croissants in the UMC staff restaurant, using a sign stating: "This croissant contains 30% fewer saturated (unhealthy) fatty acids."
Behavioral: Exchange of the basket positions of butter and margarine in the UMC staff restaurant between convenient and harder to reach locations — Exchange of the basket positions of butter and margarine in the UMC staff restaurant. In the usual (baseline) situation butter is positioned in the fridge and, therefore, less visible and harder to reach. Margarine is positioned on several convenient locations throughout the restaurant. During the two weeks intervention period these positions will be interchanged.

SUMMARY:
Rationale: Lifestyle modifications, such as increasing physical exercise and reducing dietary salt and saturated fat intake contribute to prevention of cardiovascular morbidity and mortality. Relevant improvements can already be achieved by small adaptations in everyday life. It is unclear whether simple low-cost interventions in the working environment can promote such healthy lifestyle adaptations.

Objective: To study the effect of low-cost interventions for promoting healthy lifestyle modifications.

Study design: Before-and-after intervention study. The study period will be subdivided in four parts of 2 weeks each: a run-in period, a before-measurement period, an intervention-period, and an after measurement period.

Study population: Staff and visitors of the University Medical Center Utrecht.

Study interventions:

* Promotion of stair climbing.
* Promotion of a low-salt soup alternative for the 'soup of the day'.
* Promotion of a low-fat alternative for the butter croissants.
* Exchange of the basket positions of butter and margarine between convenient and harder to reach locations.

Outcome measures:

* Number of passages through each part of the stair cases.
* Number of low-salt cream soup and normal clear soup cups sold in the hospital restaurant and ratio between them.
* Number of low-fat and normal croissants sold in the hospital restaurant and the ratio between them.
* Number of low-fat margarine servings and butter servings sold in the hospital restaurant and the ratio between them.

DETAILED DESCRIPTION:
Detailed description of the study periods:

* Run-in period: during the first 2 weeks of the study (day 1 until day 14) the baseline situation should be established and remain stable. This period is meant for study personnel to get acquainted with the study procedures.
* Before-measurement: during weeks 3 and 4 (day 15 until day 28) the measurements will start to record all endpoints and additional parameters during the baseline situation.
* Intervention-period: during weeks 5 and 6 (day 29 until day 42) the measurements will continue while the interventions are carried out.
* After measurement: during weeks 7 and 8 (day 43 until day 56) the measurements will continue while the interventions have ended and the baseline situation is restored.

ELIGIBILITY:
Dynamic population of staff and visitors of the University Medical Center Utrecht, The Netherlands

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Number of passages through each part of the stair cases | 2 weeks (including weekend days)
  Measured by wireless infrared interruption counters
Number of low-salt cream soup and normal clear soup cups sold in the hospital restaurant and ratio between them | 2 weeks (excluding weekend days)
  Assessed by the pay desk computer system administration
Number of low-fat and normal croissants sold in the hospital restaurant and the ratio between them | 2 weeks (excluding weekend days)
  Number of croissants sold will be registered on daily work sheets by the restaurant personnel
Number of low-fat margarine servings and butter servings sold in the hospital restaurant and the ratio between them | 2 weeks (excluding weekend days)
  Assessed by the pay desk computer system administration

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Dorresteijn JA, van der Graaf Y, Zheng K, Spiering W, Visseren FL. The daily 10 kcal expenditure deficit: a before-and-after study on low-cost interventions in the work environment. BMJ Open. 2013 Jan 24;3(1):e002125. doi: 10.1136/bmjopen-2012-002125. PMID 23355669